CLINICAL TRIAL: NCT06391086
Title: Neuromodulation Effect of Focused Ultrasound for Motor Recovery in Patients With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202305124DIPB
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-04

CONDITIONS: Focused Ultrasound; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with tFUS (Experimental): Treatment with tFUS
  Interventions: Device: NaviFUS® Neuronavigation-guided focused ultrasound system

INTERVENTIONS:
Device: NaviFUS® Neuronavigation-guided focused ultrasound system — The treatment protocol consists of once daily treatment for consecutive five tFUS sessions.

SUMMARY:
Transcranial focused ultrasound (tFUS) can be used as a non-invasive brain neuromodulation technique. Low-intensity focused ultrasound has been demonstrated to be safe and have neuromodulatory effects on the cerebral cortex in healthy human and animal experiments.This study aims to investigate the effect of tFUS on cortical excitability for motor recovery in patients with stroke.

DETAILED DESCRIPTION:
The study is a pilot study for feasibility, which aims to recruit 20 patients with subacute (within 3 months) stroke and unilateral hemiparesis. tFUS stimulation will be delivered. The primary outcomes are defined as cortical excitability assessment in bilateral primary motor cortex, as well as safety analysis; the secondary outcome measures include the Fugl-Meyer Assessment, Medical Research Council score, National Institutes of Health Stroke Scale (NIHSS), Barthel Index, Modified Rankin Scale and functional brain activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stroke (including hemorrhagic or ischemic stroke) diagnosed by a board-certificated physician.
* Occurrence of stroke within three months.
* Upper limb muscle strength ≤ 4 points according to the Medical Research Council Manual Muscle Testing scale.
* No previous history of stroke, epilepsy, dementia, Parkinson's disease, or other neurodegenerative diseases.
* Patients could maintain sitting posture for more than 15 minutes on a chair.
* 18 years of age or older.

Exclusion Criteria:

* History of recurrent stroke, traumatic brain injuries, brain tumors, spinal cord injury, Parkinson's disease or other musculoskeletal system diseases that may affect evaluation and treatment.
* Contraindications to focused ultrasound, including pregnancy, cardiac pacemaker or implantable medical device, abnormal connective tissue diseases, coagulopathy (PLT<100,000/μL, PT>14 seconds, APTT>36 seconds, INR>1.3), implants near or in the brain, or those deemed Unsuitable for this treatment by the physician.
* Unable to cooperate with treatment or functional assessment due to impaired consciousness or aphasia; inability to informed consent.
* Patient with cranial bone factor causing the inability of tFUS penetration.
* Patient under anticoagulants with coagulopathy (PLT<100,000/μL, PT>14 seconds, APTT>36 seconds, INR>1.3)
* Patients who are not suitable for undergoing CT imaging examination;
* Major physical illnesses and neurological disorders (such as epilepsy, brain surgery, etc.)
* Patients with metallic implants in their bodies;
* Patients taking tricyclic antidepressants, analgesics, or using antiepileptic drugs
* Individuals experiencing sleep disorders during tFUS treatment;
* Individuals with history of alcoholism
* Patients with severe or uncontrollable intracranial pressure;
* Patients requiring anticoagulants;
* Any intracranial space-occupying lesions;
* Significant calcification of intracranial vessels based on pre-treatment CT imaging;
* Subjects with lesions/wounds on the scalp in the target region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | Before treatment and on the first day (equal to day 6), first week (equal to day 12), fourth week (equal to day 33), and twelfth week (equal to day 89) after completing consecutive five tFUS sessions.
  Includes rate of minor (scalp pain, headache, short-term dizziness, nausea, vomiting, short-term weakness, short-term numbness) and severe adverse events (seizure, persistent new onset weakness, documented new intracranial hemorrhage or infarction, death)
Cortical excitability | Before treatment and on the first day (equal to day 6), first week (equal to day 12), fourth week (equal to day 33), and twelfth week (equal to day 89) after completing consecutive five tFUS sessions.
  The amplitude and latency of maximal MEP, rMT in bilateral primary motor cortex will be assessed.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity | Before treatment and on the first day (equal to day 6), first week (equal to day 12), fourth week (equal to day 33), and twelfth week (equal to day 89) after completing consecutive five tFUS sessions.
  The Fugl-Meyer Assessment for upper extremity is a standardized tool used to assess motor recovery after stroke. It consists of four items: shoulder/elbow/forearm, wrist, hand, and coordination. Each item is scored individually, with scores ranging from 0 to 2 depending on the quality of the movement. The total score ranges from 0 to 66, with higher scores indicating better motor function and recovery.
Medical Research Council score | Before treatment and on the first day (equal to day 6), first week (equal to day 12), fourth week (equal to day 33), and twelfth week (equal to day 89) after completing consecutive five tFUS sessions.
  The Medical Research Council (MRC) score is a simple and widely used scale to assess muscle strength. It rates muscle strength on a scale from 0 to 5, with 0 being no muscle contraction and 5 being normal muscle strength.
National Institutes of Health Stroke Scale (NIHSS) | Before treatment and on the first day (equal to day 6), first week (equal to day 12), fourth week (equal to day 33), and twelfth week (equal to day 89) after completing consecutive five tFUS sessions.
  The National Institutes of Health Stroke Scale (NIHSS) is a standardized tool used to assess the severity of a stroke and its effects on patients. It evaluates various neurological functions, such as consciousness, movement, sensation, and language, assigning scores ranging from 0 to 42, with higher scores indicating more severe stroke symptoms.
Barthel Index | Before treatment and on the first day (equal to day 6), first week (equal to day 12), fourth week (equal to day 33), and twelfth week (equal to day 89) after completing consecutive five tFUS sessions.
  The Barthel Index is a measure of a person's ability to perform activities of daily living. It assesses functions such as feeding, bathing, grooming, dressing, bowel and bladder control, toileting, transfers, mobility, and stairs. The score ranges from 0 to 100, with higher scores indicating greater independence.
Modified Rankin Scale | Before treatment and on the first day (equal to day 6), first week (equal to day 12), fourth week (equal to day 33), and twelfth week (equal to day 89) after completing consecutive five tFUS sessions.
  The Modified Rankin Scale is a widely used tool to assess a patient's level of disability after a stroke or other neurological disorders. It measures the degree of disability or dependence in daily activities, with scores ranging from 0 (no symptoms) to 6 (death).
Functional brain activities | Before treatment and on the first day (equal to day 6), first week (equal to day 12), fourth week (equal to day 33), and twelfth week (equal to day 89) after completing consecutive five tFUS sessions.
  Functional brain activities were detected by fNIRS (NIRSport2 NIRx Medical Technologies LLC, Glen Head, NY, USA). The subjects were requested to perform functional task (unilateral hand grasping), and brain activities was recorded by fNIRS in the following brain regions: bilateral premotor cortices, supplementary motor area, M1 and primary somatosensory cortices. The ΔHbO2 signal will be analyzed using the HOMER2 fNIRS analysis software.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ting Lin, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No